CLINICAL TRIAL: NCT00668070
Title: Protocol for a Phase II, Randomized, Double-blind, Parallel-group, Placebo-controlled, 12-week Treatment, Adaptive Proof-of-principle Study of Twice Daily Oral Dosing of a Novel PDE4 Inhibitor (ASP9831) in Subjects With Non-alcoholic Steatohepatitis (NASH)
Brief Title: A Proof-of-principle Study of Oral Treatment of Non-alcoholic Steatohepatitis With a Novel PDE4 Inhibitor ASP9831
Acronym: ASTER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9831-CL-0301; 2007-002114-19 (EudraCT Number)
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Last update posted 2013-03-21 (Estimated); Status verified 2010-11

CONDITIONS: Non-Alcoholic Steatohepatitis
Keywords: NASH; Chronic liver disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ASP9831 Low Dose (Experimental)
  Interventions: Drug: ASP9831
- ASP9831 Higher Dose (Experimental)
  Interventions: Drug: ASP9831
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP9831 — Oral
  Arms: ASP9831 Higher Dose; ASP9831 Low Dose
Drug: Placebo — Oral
  Arms: Placebo

SUMMARY:
The aim of this study is to explore the effect of a new drug (ASP9831) in patients with non-alcoholic steatohepatitis (NASH) by assessing clinical signs, laboratory data and biomarkers during a 12 week treatment period

DETAILED DESCRIPTION:
The study includes an open-label sub-study prior to the main study

ELIGIBILITY:
Inclusion Criteria:

* NASH, histologically confirmed by a liver biopsy performed within 1 year prior to first dose and randomization
* Elevated serum ALT levels

Exclusion Criteria:

* Hepatic cirrhosis
* Other known cause of liver disease
* Uncontrolled diabetes mellitis type 2, i.e. HbA1c > 8.5%
* Positive history of tuberculosis or a positive PPD skin test which is not explained by previous BCG vaccination
* History of excessive alcohol abuse within 5 years prior to screening or a current average alcohol intake of more than 20 g/day (2 units) for females or more than 30 g/day (3 units) for males
* Subject has used drugs associated with steatohepatitis within 6 months prior to screening (corticosteroids, high dose estrogens, methotrexate, amiodarone, anti-HIV drugs, tamoxifen)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2008-04; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
ALT | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Use central contact, Study Chair — Astellas Pharma Europe B.V.
Locations (27):
- Belgium (5):
  - Antwerp
  - Brussels
  - Ghent
  - La Louvière
  - Leuven
- Czechia (2):
  - Brno-Bohunice
  - Prague
- France (5):
  - Amiens
  - Angers
  - Montpellier
  - Paris
  - Pessac
- Germany (5):
  - Berlin
  - Essen
  - Frankfurt am Main
  - Mainz
  - Regensburg
- Romania (3):
  - Bucharest
  - Iași
  - Timișoara
- Switzerland (3):
  - Basel
  - Bern
  - Zurich
- United Kingdom (4):
  - Birmingham
  - London
  - Newcastle upon Tyne
  - Nottingham